CLINICAL TRIAL: NCT05097274
Title: An Imaging Study of FCH-PET-CT in Men With Prostate Cancer and a DNA Repair Gene Mutation (GENPET)
Brief Title: The GENPET Study - An Imaging Study of FCH-PET-CT in Men With Prostate Cancer and a DNA Repair Gene Mutation.
Acronym: GENPET
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR4131
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; BRCA Mutation; Mismatch Repair Gene Mutation; ATM Gene Mutation; HOXB13 Germline Mutation; CHEK2 Gene Mutation; PALB2 Gene Mutation
Keywords: FCH-PET-CT; PSMA-PET-CT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DNA repair gene mutation carriers: * Newly diagnosed with prostate cancer (any Gleason score, any stage, any PSA)
  * Biochemically progressing patients who were treated radically with surgery or radiotherapy (more than 6 months ago) and are currently not receiving hormonal treatment or chemotherapy
  * Patients on active surveillance, with a PSA doubling time of 6 months or less
  Interventions: Other: MRI pelvis or CT imaging under clinical management for Pr Ca; Other: Whole body bone scan imaging; Other: PET-CT imaging

INTERVENTIONS:
Other: MRI pelvis or CT imaging under clinical management for Pr Ca — Individuals to undergo a clinical MRI or CT scan of Pelvis and the study reviews the images.
  Other Names: Magnetic resonance imaging or computerized axial tomography
Other: Whole body bone scan imaging — bone scan of the whole body (under clinical diagnosis).
  Other Names: Bone scintigraphy
Other: PET-CT imaging — Pt will undergo a PET-CT for their clinical treatment and we will review the images of this scan.

SUMMARY:
The aim of the study is to determine if PET-CT imaging (using contrast recommended in clinical guidelines) is superior to combined bone scan and MRI/CT of the abdomen & pelvis in detecting the increased incidence of metastasis (nodal/distant outside the pelvis) in men with prostatic carcinoma with mutations in any of the following germline DNA repair genes BRCA1, BRCA2, MSH2, MSH6, MLH1, PMS2, CHEK2, PALB2, ATM.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathogenic germline mutation in any of the following genes BRCA1, BRCA2, MSH2, MSH6, MLH1, PMS2, CHEK2, PALB2 or ATM.
* Over the age of 18
* Diagnosed with prostate cancer and at a time when staging imaging is clinically indicated; either:

  * At a new diagnosis
  * Biochemically progressing patients who were treated radically with surgery or radiotherapy (more than 6 months ago) and are currently not receiving hormonal treatment or chemotherapy
  * Patients on active surveillance with a PSA doubling time of 6 months or less

Exclusion Criteria:

* Diagnosis of other malignancy (excluding basal cell cancer/squamous cell cancer of the skin) within five years of diagnosis
* Known metastatic prostate cancer, both local and distant
* Patients who have received any oncological treatment within the last six months
* Patients on any investigational drug treatment
* Patients on steroids
* Known history of inflammatory/infective diseases (e.g. sarcoidosis, tuberculosis, inflammatory bowel disease)
* Contraindications to having an MRI using the standard MRI checklist (e.g. pacemakers, aneurysm clips, claustrophobia)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient that meets the eligibility criteria and a patient at the Royal Marsden Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Sensitivity of FCH-PET-CT scan | Within 12 months of the last FCH-PET-CT scan
  To determine if the sensitivity of FCH-PET-CT is superior to combined conventional imaging (MRI (T2 and T1 weighted)/CT and bone scan) in detecting nodal and distant (outside the pelvis) metastases in BRCA1/2 germline mutation carriers with prostate cancer.

SECONDARY OUTCOMES:
2. Outline the Specificity of the FCH-PET-CT scan | Within 12 months of the last FCH-PET-CT scan
  determining the positive predictive value (PPV) and negative predictive value (NPV) in detecting metastatic disease in BRCA mutation carriers with prostate cancer
Metastasis Incidence | Within 12 months of the last FCH-PET-CT scan
  3.Incidence and sites of additional metastases identified on FCH-PET-CT compared with combined MRI/bone scan.
Impact of FCH-PET-CT findings | Within 12 months of the last FCH-PET-CT scan
  To measure the impact of FCH-PET-CT findings in changing patient management and in clinical decision making

OTHER OUTCOMES:
Incidental second primary tumours | Within 12 months of the last FCH-PET-CT scan
  To investigate the rate of incidentally detected second primary tumours in BRCA mutation carriers with prostate cancer
Prognostic significance of FCH-PET-CT findings | Within 12 months of the last FCH-PET-CT scan
  To investigate the prognostic significance of FCH-PET-CT findings (e.g. employing standard SUV parameters and heterogeneity of PET texture of the primary prostate tumour)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP FRCR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Cancer Genetics Unit, Royal Marsden Hospital, London, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be applied for via the Study Team